CLINICAL TRIAL: NCT02251964
Title: Rituximab in Life Threatening Therapy Resistant Progressive Interstitial Pneumonitis
Brief Title: Rituximab in Interstitial Pneumonitis
Acronym: RITUX-IP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Human Adams (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor-Investigator, Human Adams, Prof. Dr. D.H. Biesma, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL49534.100.14; 2013-005269-37 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Lung Diseases, Interstitial; Pneumonitis, Interstitial
Keywords: IMID; Interstitial Pneumonitis; rituximab; Immuno PET; PET/CT
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Rituximab; Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab (Other): single arm study with Zr-89-rituximab immuno PET/CT
  Interventions: Drug: Rituximab; Radiation: Zr-89-rituximab immuno PET/CT

INTERVENTIONS:
Drug: Rituximab — 2 times 1000mg dose at 14 days interval treatment
Radiation: Zr-89-rituximab immuno PET/CT — Immuno labeled PET/CT of the lungs
  Other Names: Immuno PET

SUMMARY:
This project will address rare immune mediated inflammatory diseases (IMIDs) involving the lungs, i.e. interstitial pneumonitis (IP). The main objective of this study is to assess the effects of rituximab (RTX) as a rescue therapy for progressive IMID-IP patients. The primary study parameter is pulmonary function.

The secondary objectives are to explore the application of imaging with radiolabeled RTX as early predictor for efficacy of RTX, to study the effects of RTX treatment on quality of life, and to further elucidate the pathophysiology of IMID-IP by analyzing biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the study, subjects must meet all of the following criteria:

* Age 18 to 70 years
* No previous therapy with rituximab
* At least 2 pulmonary function tests within past 6 months
* Diagnosis of co-existing IMID and a severe and / or progressive IP characterized by 3 out of the following items:
* Respiratory symptoms consistent with interstitial lung disease
* Diagnosis of usual interstitial pneumonia (UIP), non-specific interstitial pneumonia (NSIP), organizing pneumonia (OP) or a mixed form of UIP / NSIP / OP by either of the following:
* Open or video-assisted thoracic surgery (VATS) lung biopsy showing definite or probable UIP / NSIP / OP
* High Resolution Computer Tomography (HRCT) scan showing definite or probable UIP/NSIP/OP/mixed
* Forced Vital Capacity (FVC) < 50% predicted and/or diffusing capacity of the lung for carbon monoxide (DLCO) < 40% predicted or worsening of lung function as demonstrated by any one of the following within the past year:
* > 10% decrease in FVC
* > 15% decrease in DLCO
* Therapy resistance to 1st (corticosteroids) and 2nd line therapy(cyclophosphamide or azathioprine)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Residual volume >120% predicted at screening
* DLCO <25% of predicted value at screening + resting Oxygen Saturation (SAO2) without external oxygen <90%
* History of unstable or deteriorating cardiac or neurological disease
* Pregnancy or lactation
* Hematology lower than specified limits (leucocytes)
* Positive HIV, hepatitis B or C serology
* Pre-existing conditions which lead to a life expectancy of less than 6 months
* Receipt of any vaccine, particularly live viral vaccines, within 4 weeks before first rituximab dose
* Hypersensitivity for murine proteins

NOTE:

* Fever (>37,9 °C) at presentation is reason to delay therapy by 1 week
* Evidence of active infection is reason to postpone rituximab treatment until no further signs of active infection
* Severe renal impairment is not a contraindication for rituximab therapy, however, if patients (might) require dialysis frequently they will be excluded from the study group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary function (VC, DLCO) | 6 - 12 months
  establish a change from the downward decline in pulmonary function (absolute values and values predicted of VC = Vital Capacity and DLCO = Diffusion capacity of Lung Carbon monoxide)

SECONDARY OUTCOMES:
Zr-89 Immuno PET | 3, 6 days after injection
  This is a scan with radiolabelled rituximab (visualizing rituximab activity in the lungs). Calculated activity (SUV) in the lungs vs. blood pool vs liver vs.control group (n=15) is measured with standard deviation. The amount of uptake in the lungs and the clinical response of patients will be correlated to determine a correlation.

CONTACTS AND LOCATIONS:
Overall Officials: J C Grutters, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Derived] Adams H, van de Garde EMW, Vugts DJ, Grutters JC, Oyen WJG, Keijsers RG. [89Zr]-immuno-PET prediction of response to rituximab treatment in patients with therapy refractory interstitial pneumonitis: a phase 2 trial. Eur J Nucl Med Mol Imaging. 2023 Jun;50(7):1929-1939. doi: 10.1007/s00259-023-06143-1. Epub 2023 Feb 24. PMID 36826476